CLINICAL TRIAL: NCT05513937
Title: Open-laBel, Multicenter, multinatiOnal, inTerventional Clinical Trial to Assess effIcacy and Safety of the Extemporaneous Combination of nEbivoLol and amLodipine in Grade 1-2 Hypertensive patIents Versus Each Monotherapy
Brief Title: Effectiveness and Safety of Combination of Nebivolol and Amlodipine in Hypertensive Patients Versus Each Monotherapy
Acronym: Botticelli
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Menarini International Operations Luxembourg SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MEIN/21/AmNe-Hyp/001
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Results first posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Nebivolol; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nebivolol 5 mg (Active Comparator): MONOTHERAPY PHASE 4 weeks (Run-in from -4 week to week 0):
  patients will be treated with Nebivolol 5mg
  COMBINATION THERAPY PHASE 8 weeks (from week 0 to week 8):
  uncontrolled patients during Monotherapy Phase will be treated with the extemporaneous combination of Nebivolol 5mg and Amlodipine 5mg for 4 weeks (from week 0 to week 4). Amlodipine 10mg will replace Amlodipine 5mg in uncontrolled patients for further 4 weeks (from week 4 to week 8) while controlled patients with Nebivolol 5mg/Amlodipine 5mg will continue with the same therapy.
  Interventions: Drug: Nebivolol; Drug: Amlodipine
- Amlodipine 5/10 mg (Active Comparator): MONOTHERAPY PHASE 4 weeks (Run-in from -4 week to week 0):
  patients will be treated with Amlodipine 5mg
  COMBINATION THERAPY PHASE 8 weeks (from week 0 to week 8):
  uncontrolled patients during Monotherapy Phase will be treated with the extemporaneous combination of Nebivolol 5mg and Amlodipine 5mg for 4 weeks (from week 0 to week 4). Amlodipine 10mg will replace Amlodipine 5mg in uncontrolled patients for further 4 weeks (from week 4 to week 8) while controlled patients with Nebivolol 5mg/Amlodipine 5mg will continue with the same therapy.
  Interventions: Drug: Nebivolol; Drug: Amlodipine

INTERVENTIONS:
Drug: Nebivolol — Tablets administered orally once daily according instructions provided by Principal Investigator.
Drug: Amlodipine — Tablets of 5mg and 10mg administered orally once daily according instructions provided by Principal Investigator.

SUMMARY:
Study to assess the anti-hypertensive efficacy and safety of the extemporaneous combination of Nebivolol 5 mg in combination with Amlodipine 5 mg or AML 10 mg in lowering the sitting diastolic BP after 8 weeks of treatment inpatients with uncontrolled BP previously treated with Nebivolol (NEB) or Amlodipine (5 mg) monotherapies for at least 4 weeks.

DETAILED DESCRIPTION:
Approximately 290 patients are planned to be screened to ensure at least 216 patients complete the run-in period and start with the assessment period.

Grade 1 - 2 hypertensive patients [BP ranging from ≥140 to ≤179 mmHg for Systolic Blood Pressure (SBP) and from ≥90 to ≤109 mmHg for Diastolic Blood Pressure (DBP)] on treatment with any Beta Blocker (BB) or Calcium Channel Blocker (CCB), including NEB (only 5 mg dosage allowed) or AML (only 5 mg dosage allowed) for at least one month prior to Visit 1 will be screened for eligibility.

Allowed CCBs at screening includes Felodipine, isradipine, lacidipine, lercanidipine, nicardipine, nifedipine, and nisoldipine. Patients treated with Amlodipine or Nebivolol in dosages higher than 5 mg/daily will not be eligible.

On the same day of the Screening visit, the eligible patients will enter into a run-in period of 4 weeks after screening, during which:

* Patients receiving NEB 5 mg or AML 5 mg will continue the same therapy for 4 weeks.
* Patients on any other BBs or CCBs will be switched to NEB 5 mg or AML 5 mg. Patients entering this phase in therapy with NEB 5 mg or AML 5 mg should be in a 1:1 ratio.

After 4 weeks (±2 days) of run-in period of monotherapy, the BP will be further assessed (Visit 2). Patients with uncontrolled BP levels (sitting SBP/DBP ≥130/80 mmHg) at Visit 2, with the treatment adherence (ranging between 80% to 120%) and who did tolerate the treatment will enter into the assessment period and will be assigned to the extemporaneous combination of NEB 5 mg and AML 5 mg. Patients with controlled BP levels (sitting SBP/DBP <130/80 mmHg) and/or who do not tolerate the treatment or have an adherence range below 80% or above 120%, will be withdrawn from the study.

After 4 weeks ±2 days in the assessment period, patients BP will be further evaluated at Visit 3: patients with controlled BP levels (sitting SBP/DBP <130/80 mmHg) will continue the same extemporaneous combination, while patients with uncontrolled BP levels will be uptitrated from extemporaneous combination NEB/AML 5/5 mg to extemporaneous combination of NEB/AML 5/10 mg for further 4 weeks.

At the end of the assessment period (8 weeks ±4 days), the patients will attend an End of Treatment Visit 4.

To correctly evaluate the additional effect of the combination therapy, the number of patients with uncontrolled BP on NEB or AML monotherapy needs to be balanced at Visit 2. In order to maintain a 1:1 ratio during the assessment period, a cap of 110 patients for each treatment arm (ie. NEB and AML) will be included at Visit 2 in order to maintain a balanced number of uncontrolled patients entering the assessment period for each drug. The evaluation will be done every 50 patients. If the rate of entrance in the assessment period for one of the 2 tested drugs will deviate more than 5%, a corrective measure will be initiated.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients with Grade 1 - 2 hypertension with mean sitting SBP ≥140 mmHg and ≤179 mmHg and/or mean sitting DBP ≥90 mmHg and ≤109 mmHg at screening (in accordance with the 2018 European Society of Cardiology / European Society of Hypertension guidelines definition), ≥18 and <65 years of age, on monotherapy treatment either with BBs or CCBs for at least 4 weeks before Visit 1 (screening).
2. Patients are able to understand and have freely given written informed consent at Screening Visit.
3. Patients who are able to comply with all study procedures and who are available for the duration of the study.
4. Ability to take oral medication and willing to adhere to the drug regimen.
5. Female patients are eligible to participate if not pregnant, or not breastfeeding and if they refrain from donating or storing eggs. For females of reproductive potential: use of highly effective contraception (eg. method of birth control throughout the study period and for 4 weeks after study completion defined as a method which results in a failure rate of <1% per year) such as:

   * Combined hormonal contraception (estrogen- and progestogen-containing) associated with inhibition of ovulation (oral, intravaginal, and transdermal).
   * Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, and implantable).
   * Intrauterine device.
   * Intrauterine hormone-releasing system.
   * Bilateral tubal occlusion.
   * Vasectomized partner (procedure conducted at least 2 months before the screening), (provided the partner is the sole sexual partner of the trial participant and that the vasectomized partner has received medical assessment of the surgical success).
6. A male patient must agree to use contraception during the whole study period and for at least 1 week after the last dose of study treatment and refrain from donating sperms during this period.

Exclusion Criteria:

1. Patients with significant history of hypersensitivity to nebivolol, amlodipine, other BBs or other dihydropyridines, or any related products (including excipients of the formulations) as outlined in the relevant Investigators Brochures, summary of product characteristics12,13 or local package inserts for NEB and AML.
2. Patients with serious disorders (in the opinion of the Investigator) which may limit the ability to evaluate the efficacy or safety of the tested medications, including cerebrovascular, cardiovascular, renal, respiratory, hepatic, gastrointestinal, endocrine or metabolic, hematological, or oncological, neurological, and psychiatric diseases. The same applies for immunocompromised and/or neutropenic patients.
3. Patients having a history of the following conditions within the last 6 months: myocardial infarction, unstable angina pectoris, percutaneous coronary intervention, bypass surgery, heart failure, hypertensive encephalopathy, valve replacement (transcatheter aortic valve implantation, mitraclip), cerebrovascular accident (stroke), or transient ischemic attack.
4. Patients with condition of hypotension with SBP <90 mmHg and/or DBP <60 mmHg.
5. Acute heart failure, cardiogenic shock, or episodes of heart failure decompensation requiring intravenous inotropic therapy.
6. Patients with secondary hypertension of any etiology including renal diseases, pheochromocytoma, Cushing's syndrome, hyperaldosteronism, renovascular disease, and thyroid disorders.
7. Patients with a narrowing of the aortic or bicuspid valve, an obstruction of cardiac outflow (obstructive, hypertrophic cardiomyopathy), obstruction of the outflow tract of the left ventricle (eg. high grade aortic stenosis) or symptomatic coronary disease.
8. Patients with severe renal impairment or renal transplant.
9. Patients with clinically relevant hepatic impairment.
10. Patients with sick sinus syndrome, including sino-atrial block.
11. Patients with second- or third-degree heart block (without a pacemaker).
12. Patients with history of bronchospasm and bronchial asthma.
13. Patients with untreated pheochromocytoma.
14. Patients with bradycardia (heart rate <60 bpm; <50 bpm in patients already on BBs treatment).
15. Patient with metabolic acidosis.
16. Patients with severe peripheral circulatory disturbances.
17. Participation in another interventional study within the last 4 weeks before Screening Visit (Visit 1).
18. Patients with diseases that, in the opinion of the Investigator, prevent a careful adherence to the protocol.
19. Patients using and not suitable for withdrawing the prohibited medications prior to the administration of study treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Volpe, Principal Investigator — University "Sapienza" Rome
Locations (1):
- Medical Center Hera EOOD, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: MONOTHERAPY PERIOD:Patients are treated with NEB 5 mg or AML 5 mg during the Run in period (week -4 to week 0) according the assigned arms. Uncontrolled patients enter the COMBINATION THERAPY PERIOD, a one arm assessment period of 8 weeks (week 0 to week 8), where patient are treated with extemporaneous combination of NEB 5 mg/AML 5mg for 4 weeks. AML 10mg will replace AML 5mg in uncontrolled patients for further 4 weeks while controlled patients will continue with the same combination therapy.
Groups:
- Run-In Nebivolol 5mg: MONOTHERAPY PHASE (Run-in 4 weeks from -4 week to week 0):
  patients will be treated with Nebivolol 5mg Nebivolol: Tablets administered orally once daily according instructions provided by Principal Investigator.
- Run-In Amlodipine 5mg: MONOTHERAPY PHASE (Run-in 4 weeks from -4 week to week 0):
  patients will be treated with Amlodipine 5mg. Amlodipine: Tablets of 5mg administered orally once daily according instructions provided by Principal Investigator.
- Combination Therapy Nebivolol 5mg/ Amlodipine 5mg: COMBINATION THERAPY PHASE (8 weeks from week 0 to week 8):
  uncontrolled patients taking Nebivolol 5 mg or Amlodipine 5mg during the respective Run-in Phases, will be treated with the extemporaneous combination of Nebivolol 5mg and Amlodipine 5mg for 4 weeks (from week 0 to week 4).Amlodipine 10mg will replace Amlodipine 5mg in uncontrolled patients for further 4 weeks (from week 4 to week 8) while controlled patients with Nebivolol 5mg/Amlodipine 5mg will continue with the same therapy.
  Nebivolol: Tablets administered orally once daily according instructions provided by Principal Investigator.
  Amlodipine: Tablets of 5mg administered orally once daily according instructions provided by Principal Investigator.
- Combination Therapy Nebivolol 5mg/ Amlodipine 10mg: COMBINATION THERAPY PHASE (4 weeks from week 4 to week 8):
  Amlodipine 10mg will replace Amlodipine 5mg in uncontrolled patients treated with the extemporaneous combination of Nebivolol 5mg and Amlodipine 5mg for 4 weeks (from week 0 to week 4), for further 4 weeks (from week 4 to week 8) while controlled patients with Nebivolol 5mg/Amlodipine 5mg will continue with the same therapy.
  Nebivolol: Tablets administered orally once daily according instructions provided by Principal Investigator.
  Amlodipine: Tablets of 10mg administered orally once daily according instructions provided by Principal Investigator.
Period: Run in (-4 Week to 0) Monotherapy Phase
Arm/Group | Run-In Nebivolol 5mg | Run-In Amlodipine 5mg | Combination Therapy Nebivolol 5mg/ Amlodipine 5mg | Combination Therapy Nebivolol 5mg/ Amlodipine 10mg
Started | 143 | 158 | 0 | 0
Completed | 139 | 152 | 0 | 0
Not Completed | 4 | 6 | 0 | 0
Not completed — Newly developed or not previously recognized exclusion criteria | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 2 | 5 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: Combination Therapy (0 to 4 Weeks)
Arm/Group | Run-In Nebivolol 5mg | Run-In Amlodipine 5mg | Combination Therapy Nebivolol 5mg/ Amlodipine 5mg | Combination Therapy Nebivolol 5mg/ Amlodipine 10mg
Started | 0 | 0 | 279 | 0
Completed | 0 | 0 | 279 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Combination Therapy (4 to 8 Weeks)
Arm/Group | Run-In Nebivolol 5mg | Run-In Amlodipine 5mg | Combination Therapy Nebivolol 5mg/ Amlodipine 5mg | Combination Therapy Nebivolol 5mg/ Amlodipine 10mg
Started | 0 | 0 | 185 (185 are patients that have maintained Neb 5/Aml 5 mg during all the assessment period (COMBINATION THERAPY PERIOD) from week 0 to week 8) | 94 (94 are patients that started the assessment period (COMBINATION THERAPY PERIOD) with Neb 5mg/Aml 5mg and, at week 4,were uptitrated to Neb 5mg/Aml 10mg)
Completed | 0 | 0 | 182 (182 are patients that have completed combination therapy with Nebivolol 5mg and Amlodipine 5mg) | 94 (94 are patients that have completed combination therapy with Nebivolol 5mg and Amlodipine 10mg)
Not Completed | 0 | 0 | 3 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Combination Therapy Nebivolol 5mg/ Amlodipine 5mg: COMBINATION THERAPY PHASE (8 weeks from week 0 to week 8):
  uncontrolled patients taking Nebivolol 5 mg or Amlodipine 5mg during the respective Run-in Phases, will be treated with the extemporaneous combination of Nebivolol 5mg and Amlodipine 5mg for 4 weeks (from week 0 to week 4). Amlodipine 10mg will replace Amlodipine 5mg in uncontrolled patients for further 4 weeks (from week 4 to week 8) while controlled patients with Nebivolol 5mg/Amlodipine 5mg will continue with the same therapy.
  Nebivolol: Tablets administered orally once daily according instructions provided by Principal Investigator.
  Amlodipine: Tablets of 5mg administered orally once daily according instructions provided by Principal Investigator.
- Combination Therapy Nebivolol 5mg/ Amlodipine 10mg: COMBINATION THERAPY PERIOD: (4 weeks from Week 4 to Week 8):
  Amlodipine 10mg will replace Amlodipine 5mg in uncontrolled patients treated with the extemporaneous combination of Nebivolol 5mg and Amlodipine 5mg for 4 weeks (from Week 0 to Week 4), for further 4 weeks, while controlled patients with Nebivolol 5mg/Amlodipine 5mg, will continue with the same therapy.
  Nebivolol: Tablets administered orally once daily according instructions provided by Principal Investigator.
  Amlodipine: Tablets of 5mg and 10mg administered orally once daily according instructions provided by Principal Investigator.
- Total: Total of all reporting groups
Arm/Group | Combination Therapy Nebivolol 5mg/ Amlodipine 5mg | Combination Therapy Nebivolol 5mg/ Amlodipine 10mg | Total
Number analyzed (Participants) | 185 | 94 | 279
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (8.14) | 53.4 (8.02) | 52.2 (8.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 45 | 144
  Male | 86 | 49 | 135
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 185 | 94 | 279
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Sitting Diastolic Blood Pressure (DBP) Between Visit 2 (Week 0) and Visit 4 (Week 8)
Description: To assess the antihypertensive efficacy of the extemporaneous combination of Nebivolol (NEB) 5 mg in combination with Amlodipine (AML) 5 mg or AML 10 mg in lowering the sitting diastolic BP between Visit 2 (Week 0) and Visit 4 (Week 8) in patients with uncontrolled BP previously treated with Nebivolol or Amlodipine (5 mg) monotherapies for at least 4 weeks during run-in period.
Time Frame: From Visit 2 (week 0) to Visit 4 (week 8) for a total of 8 weeks
Population: Primary endpoint (as per protocol assessed in patients who received combination therapy regardless of AML dose), is defined as mean difference in sitting diastolic blood pressure between Visit 2 (Week 0, Baseline Visit of the combination therapy) and Visit 4 (Week 8, End of Study Visit). This is not a comparison of two different arms, but a comparison of two measurements taken from the same patient treated with combination therapy (single arm paired pre- vs. post-combination therapy comparison)
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Combination Therapy Phase Nebivolol 5mg/Amlodipine 5 or 10 mg: Combination Therapy Phase (8 weeks) from Visit 2 (week 0) to Visit 4 (week 8): uncontrolled patients with Monotherapy (Nebivolol 5 mg or Amlodipine 5 mg) are treated with the extemporaneous combination of Nebivolol 5 mg and Amlodipine 5mg for 4 weeks. Amlodipine 10mg will replace Amlodipine 5mg in uncontrolled patients for further 4 weeks while controlled patients with Nebivolol 5mg/Amlodipine 5mg will continue with the same therapy.
  Nebivolol: Tablets administered orally once daily according instructions provided by Principal Investigator.
  Amlodipine: Tablets of 5mg and 10mg administered orally once daily according instructions provided by Principal Investigator.
Arm/Group | Combination Therapy Phase Nebivolol 5mg/Amlodipine 5 or 10 mg
Number analyzed (Participants) | 276
mmHg | -15.2 (8.32)
Statistical Analysis 1: Comparison: Combination Therapy Phase Nebivolol 5mg/Amlodipine 5 or 10 mg; Test type: Superiority; p < 0.001, Wilcoxon signed rank test; Mean difference pre vs post = -15.2, Standard Deviation 8.32

ADVERSE EVENTS:
Time Frame: From Informed Consent signature at screening visit (Visit 1) occurring 4 week previous than Baseline assessment (Week 0 - Visit 2) to last visit at Week 8 (Visit 4) for an average of 12 weeks. Furthermore patients having any ongoing Adverse Event/Serious Adverse Event at the end of the treatment (Week 8 - Visit 4), will be followed for further 2 weeks via a phone call to check about the status of the Adverse Events/Serious Adverse Events, extending the time frame to a total of 14 weeks.
Description: Safety analyses were carried out using the Safety analysis population, which was defined as all patients in the Enrolled population who received at least one dose of study medication (i.e., monotherapy and/or combination therapy )
  If a patient reports the same Adverse Event (AE) more than once within that System Organ Class/Preferred Term, then that patient will be counted only once for that System Organ Class or Preferred Term
Groups:
- Nebivolo 5 mg MONOTHERAPY PERIOD: All patients Enrolled who received at least one dose of Nebivolol 5mg in Monotherapy during the Run in Phase ( from -4 week to week 0)
- Amlodipine 5 mg MONOTHERAPY PERIOD: All patients Enrolled who received at least one dose of Amlodipine 5mg in Monotherapy during the Run in Phase ( from -4 week to week 0)
- Nebivolo 5mg/Amlodipine 5 mg COMBINATION THERAPY PERIOD: All patients Enrolled who received at least one dose of the Combination therapy: Nebivolol 5mg/Amlodipine 5 from week 0 to week 8
- Nebivolo 5mg/Amlodipine 10mg COMBINATION THERAPY PERIOD: All patients Enrolled who received at least one dose of the Combination therapy: Nebivolol 5mg/Amlodipine 10mg from week 0 to week 8
Arm/Group | Nebivolo 5 mg MONOTHERAPY PERIOD | Amlodipine 5 mg MONOTHERAPY PERIOD | Nebivolo 5mg/Amlodipine 5 mg COMBINATION THERAPY PERIOD | Nebivolo 5mg/Amlodipine 10mg COMBINATION THERAPY PERIOD
All-Cause Mortality (participants affected / at risk) | 0/143 | 0/158 | 0/279 | 0/94
Serious Adverse Events (participants affected / at risk) | 0/143 | 0/158 | 0/279 | 0/94
Other Adverse Events (participants affected / at risk) | 4/143 | 2/158 | 35/279 | 9/94
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nebivolo 5 mg MONOTHERAPY PERIOD (N=143) | Amlodipine 5 mg MONOTHERAPY PERIOD (N=158) | Nebivolo 5mg/Amlodipine 5 mg COMBINATION THERAPY PERIOD (N=279) | Nebivolo 5mg/Amlodipine 10mg COMBINATION THERAPY PERIOD (N=94)
Flushing (Vascular disorders) | 0 | 0 | 1 | 0
Feeling Hot (General disorders) | 0 | 0 | 1 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 2 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 1 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 1 | 0
Heart rate increased (Investigations) | 0 | 0 | 1 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 3
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 7 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 3 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Peripheral swelling (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Thyroid disorder (Endocrine disorders) | 0 | 1 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 3
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-09-27): https://cdn.clinicaltrials.gov/large-docs/37/NCT05513937/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-23): https://cdn.clinicaltrials.gov/large-docs/37/NCT05513937/SAP_001.pdf